CLINICAL TRIAL: NCT04405336
Title: Effect of Tab Block and Patient Controlled Analgesia in Cesarean Section
Brief Title: Tab Block and Patient Controlled Analgesia in CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: tab block
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- giving tab block (Active Comparator): giving patients tab block
  Interventions: Drug: tab block; Drug: women who will not receive tab block or PCA
- giving PCA (Active Comparator): Giving PCA to patients
  Interventions: Drug: PCA; Drug: women who will not receive tab block or PCA
- Patients who will not receive PCA or tab block (No Intervention): No tab block or PCA

INTERVENTIONS:
Drug: tab block — injection of tab block to women who are doing cs
  Arms: giving tab block
Drug: PCA — giving women PCA
  Arms: giving PCA
Drug: women who will not receive tab block or PCA — no tab block or PCA will be given
  Arms: giving PCA; giving tab block

SUMMARY:
cesarean section rate become increasing nowadays

DETAILED DESCRIPTION:
indication of cesarean section are different from case to case and the use of pain controlling agents is very important to relieve post operative pain

ELIGIBILITY:
Inclusion Criteria:

* women coming for an elective CS

Exclusion Criteria:

* women who has a n emergency CS or complicated normal deivery needs urgent CS

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women undergoing CS
Enrollment: 140 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
The number of women who will feel less pain post CS | 2 days
  the degree of pain that will be felt post CS

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt